CLINICAL TRIAL: NCT06848374
Title: Dose Comparison for the Treatment of Adhesive Capsulitis with Hydrodilatation and Corticosteroid Using an Anterior Approach Under Ultrasound-Guidance
Brief Title: Dose Efficacy in Adhesive Capsulitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Nimish Mittal, Assistant Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-5123
Record Dates: First submitted 2025-02-08; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Adhesive Capsulitis of the Shoulder
Keywords: Frozen shoulder; hydrodilatation
MeSH Terms: conditions — Bursitis | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 40mg methylprednisolone dose
  Interventions: Drug: 40 mg Methylprednisolone
- Group B (Active Comparator): 80mg methylprednisolone dose
  Interventions: Drug: 80 mg Methylprednisolone

INTERVENTIONS:
Drug: 40 mg Methylprednisolone — Ultrasound guided injection of 40mg methylprednisolone injection
  Arms: Group A
Drug: 80 mg Methylprednisolone — Ultrasound guided injection of 40mg methylprednisolone injection
  Arms: Group B

SUMMARY:
The purpose of this study is to find out if the treatment of adhesive capsulitis with 40 mg of methylprednisolone in combination with a hydrodilatation is comparable to 80 mg of methylprednisolone for pain reduction, improving shoulder mobility, and reducing side effects.

Researchers will enroll 40 people in this study which is taking place solely at the Toronto Rehabilitation Institute, University Avenue. This study should take approximately 12 months to complete and the results should be known in about 15 to 18 months. During this study, patients will receive an ultrasound guided shoulder hydrodilatation combined with corticosteroid after "randomized" into one of the groups (40 mg vs 80 mg). This is a double blind study as both patients and physicians would not know the group patient was randomized to.

Pain scores, Range of Motion and few other questionnaires wold be completed to track the response to the interventions at baseline prior to injection, four weeks after the procedure and 3 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnostic of adhesive capsulitis of the shoulder

Exclusion Criteria:

* Injection received in the affected shoulder < 3 months ago (any kind)
* History of previous surgery in the affected shoulder
* Glenohumeral osteoarthritis more than mild on the xray
* Pregnancy
* Blood thinner (other than Aspirin 80 mg) or bleeding disorder
* Active infection (requiring antibiotic)
* Allergy to steroid or lidocaine
* Cognitive impairment
* Active litigation
* Inflammatory connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale | 3 months
  Change in pain scores using Numeric Pain Rating scale form baseline to 3 months

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index score | 3 months
  change in pain scores using Shoulder Pain and Disability Index score form baseline to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabilitation Institution, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No